CLINICAL TRIAL: NCT00746278
Title: A Random Clinical Trial of the Impact of Electrocoagulation on Ovarian Reserve After Laparoscopic Excision of Ovarian Cyst
Brief Title: A Random Clinical Trial (RCT) of the Impact of Electrocoagulation on Ovarian Reserve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Shandong University (Other)
Responsible Party: Xiayong Wang Ph.D, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPH-CL-080512
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2008-05

CONDITIONS: Ovarian Cyst
Keywords: Ovarian Cysts; Electrocoagulation; Ovarian Function Tests; Laparoscopy
MeSH Terms: conditions — Ovarian Cysts; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Laparoscopic ovarian cystectomy using bipolar
  Interventions: Procedure: Laparoscopic ovarian cystectomy using bipolar
- 2 (Experimental): Laparoscopic ovarian cystectomy using ultrasonic scalpel electrocoagulation
  Interventions: Procedure: Laparoscopic ovarian cystectomy using ultrasonic scalpel
- 3 (Active Comparator): Laparoscopic ovarian cystectomy using suture
  Interventions: Procedure: Laparoscopic ovarian cystectomy using suture

INTERVENTIONS:
Procedure: Laparoscopic ovarian cystectomy using bipolar — Laparoscopic ovarian cystectomy using bipolar
  Arms: 1
Procedure: Laparoscopic ovarian cystectomy using ultrasonic scalpel — Laparoscopic ovarian cystectomy using ultrasonic scalpel
  Arms: 2
Procedure: Laparoscopic ovarian cystectomy using suture — Laparoscopic ovarian cystectomy using suture
  Arms: 3

SUMMARY:
Laparoscopic ovarian cystectomy is widely used for the removal of benign ovarian cysts but damage to ovarian reserve caused by electrocoagulation has recently been questioned.

The purpose of this study is to investigate the impact of bipolar and ultrasonic scalpel electrocoagulation on ovarian reserve after laparoscopic excision of ovarian cyst.

DETAILED DESCRIPTION:
Laparoscopic ovarian cystectomy is currently considered the treatment of choice in women with benign ovarian cyst and has gained increasing acceptance among gynecological surgeons(1). However, the safety of this technique in terms of ovarian damage to the operated gonad caused by electrocoagulation has recently been questioned. Many evidences support that the removal of ovarian cysts is associated with an injury to ovarian reserve. On the contrary, some retrospective studies did not show adverse outcomes compared with the control group (tubal infertility) . There is a lack of good clinical and scientific evidence such as randomized controlled study to report definitively the impact of electrocoagulation on ovarian reserve after laparoscopic excision of ovarian cyst.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years
* ultrasound diagnosis as unilateral ovarian cyst and the average size between 5cm and 10cm
* no clinical and sonographic suspicion of ovarian cancer
* regular menstrual cycles defined as cycle length between 25 and 35 days in the 6 months before surgery
* sonographic normal contralateral ovary
* agreement to be enrolled in the study.

Exclusion Criteria:

* prior ovarian surgery or known endocrine disease
* surgical necessity to perform adnexectomy
* intraoperative diagnosis of an abnormal contralateral ovary
* post operative pathologic diagnosis was not benign ovarian cyst
* oral contraceptive use before surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Serum FSH and inhibin-B and Anti-Mullerian hormone(AMH) assays | 12 months

SECONDARY OUTCOMES:
Transvaginal ultrasound examinations for basal antral follicle number, mean ovarian diameter and peak systolic velocity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Zhong Li,, M.D.Ph.D., Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

REFERENCES:
- [Background] Candiani M, Barbieri M, Bottani B, Bertulessi C, Vignali M, Agnoli B, Somigliana E, Busacca M. Ovarian recovery after laparoscopic enucleation of ovarian cysts: insights from echographic short-term postsurgical follow-up. J Minim Invasive Gynecol. 2005 Sep-Oct;12(5):409-14. doi: 10.1016/j.jmig.2005.06.006. PMID 16213426
- [Background] Ho HY, Lee RK, Hwu YM, Lin MH, Su JT, Tsai YC. Poor response of ovaries with endometrioma previously treated with cystectomy to controlled ovarian hyperstimulation. J Assist Reprod Genet. 2002 Nov;19(11):507-11. doi: 10.1023/a:1020970417778. PMID 12484492
- [Background] Loh FH, Tan AT, Kumar J, Ng SC. Ovarian response after laparoscopic ovarian cystectomy for endometriotic cysts in 132 monitored cycles. Fertil Steril. 1999 Aug;72(2):316-21. doi: 10.1016/s0015-0282(99)00207-1. PMID 10439003
- [Background] Nargund G, Cheng WC, Parsons J. The impact of ovarian cystectomy on ovarian response to stimulation during in-vitro fertilization cycles. Hum Reprod. 1996 Jan;11(1):81-3. doi: 10.1093/oxfordjournals.humrep.a019043. PMID 8671163
- [Background] Somigliana E, Ragni G, Benedetti F, Borroni R, Vegetti W, Crosignani PG. Does laparoscopic excision of endometriotic ovarian cysts significantly affect ovarian reserve? Insights from IVF cycles. Hum Reprod. 2003 Nov;18(11):2450-3. doi: 10.1093/humrep/deg432. PMID 14585900